CLINICAL TRIAL: NCT04004975
Title: Phase II Clinical Trials on Anlotinib for the Treatment of Recurrent Glioblastoma.
Brief Title: Clinical Study on the Treatment of Recurrent Glioblastoma With Anlotinib
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Rongjie Tao, Chief Physician, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ShandongCHI006
Record Dates: First submitted 2019-07-01; First posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Recurrent Glioblastoma
Keywords: anlotinib Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — anlotinib

STUDY DESIGN:
Intervention Model Description: one-armed controlled clinical trial
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- anlotinib (Experimental): 12 mg daily from day 1 to 14 of a 21-day cycle
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — Anlotinib is a multitarget receptor tyrosine kinase inhibitor which inhibits vascular endothelial growth factor receptor (VEGFR) 1-3, fibroblast growth factor receptor (FGFR) 1-4, platelet-derived growth factor receptors (PDGFR) α/β, c-Kit, and Met.
  Other Names: Fu Ke Wei

SUMMARY:
Anlotinib is a novel small molecule multi-target tyrosine kinase inhibitor that can inhibit tumor angiogenesis and inhibit tumor cell growth. We performed second-generation gene sequencing on pathological specimens and cerebrospinal fluid of patients with recurrent glioblastoma.If patients have a genetic mutation （VEGFR，Kit，PDGFR，FGFR）and meet other eligibility criteria, they will be treated with antroinib. The initial observation targets were progression-free survival and adverse reactions. The secondary objective was overal survival.

DETAILED DESCRIPTION:
INCLUSION CRITERIA:

1. Histologically confirmed World Health Organization (WHO) Grade IV glioblastoma.;
2. Radiographic evidence of tumour progression or recurrence;
3. The second-generation gene sequencing on pathological specimens and cerebrospinal fluid show at least one genetic mutation of the four genes (VEGFR，Kit，PDGFR，FGFR);
4. ≥ 18 years of age;
5. Karnofsky performance status (KPS) ≥ 70;
6. Corticosteroid dose must be stable or decreasing for at least 5 days prior to the scan.
7. a new baseline scan is required 1.7 Measurable disease as per Response Assessment in Neuro-Oncology (RANO) criteria;
8. Estimated survival of at least 3 months;
9. signed informed consent form;
10. Hgb > 9 gm; absolute neutrophil count (ANC) > 1500/μl; platelets > 100,000; Creatinine < 1.5 times the upper limit of laboratory normal value; Bilirubin < 2 times the upper limit of laboratory normal value; serum glutamate pyruvate transaminase (SGPT) or serum glutamate oxaloacetate transaminase (SGOT) < 3 times the upper limit of laboratory normal value;

EXCLUSION CRITERIA:

Exclusion Criteria:

1. Subjects with newly diagnosed GBM
2. Pregnant women or nursing mothers cannot participate in the study. Women of childbearing age must have a negative pregnancy test within 72 hours prior to study entry. Women of childbearing potential must practice medically approved contraceptive precautions;
3. Abnormal hematological results at inclusion with: Neutrophils < 1,500/mm3; Blood-platelets < 100,000/mm3
4. Severe or chronic renal insufficiency (creatinine clearance ≤ 30 ml/min);
5. Patient unable to follow procedures, visits, examinations described in the study;
6. Any usual formal indication against imaging examinations (important claustrophobia, pacemaker);

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed World Health Organization (WHO) Grade IV glioblastoma.;
2. Radiographic evidence of tumour progression or recurrence;
3. The second-generation gene sequencing on pathological specimens and cerebrospinal fluid show at least one genetic mutation of the four genes (VEGFR，Kit，PDGFR，FGFR);
4. ≥ 18 years of age;
5. Karnofsky performance status (KPS) ≥ 70;
6. Corticosteroid dose must be stable or decreasing for at least 5 days prior to the scan.
7. a new baseline scan is required 1.7 Measurable disease as per Response Assessment in Neuro-Oncology (RANO) criteria;
8. Estimated survival of at least 3 months;
9. signed informed consent form;
10. Hgb > 9 gm; absolute neutrophil count (ANC) > 1500/μl; platelets > 100,000; Creatinine < 1.5 times the upper limit of laboratory normal value; Bilirubin < 2 times the upper limit of laboratory normal value; serum glutamate pyruvate transaminase (SGPT) or serum glutamate oxaloacetate transaminase (SGOT) < 3 times the upper limit of laboratory normal value;

Exclusion Criteria:

1. Subjects with newly diagnosed GBM
2. Pregnant women or nursing mothers cannot participate in the study. Women of childbearing age must have a negative pregnancy test within 72 hours prior to study entry. Women of childbearing potential must practice medically approved contraceptive precautions;
3. Abnormal hematological results at inclusion with: Neutrophils < 1,500/mm3; Blood-platelets < 100,000/mm3
4. Severe or chronic renal insufficiency (creatinine clearance ≤ 30 ml/min);
5. Patient unable to follow procedures, visits, examinations described in the study;
6. Any usual formal indication against imaging examinations (important claustrophobia, pacemaker);

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-06-25 (Estimated); Primary Completion 2020-07-25 (Estimated); Study Completion 2021-07-25 (Estimated)

PRIMARY OUTCOMES:
Progress free survival (PFS) | each 42 days up to PD or death(up to 24 months)
  PFS defined as the time from first dose of study treatment until the first date of either objective disease progression or death due to any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | From randomization until death (up to 24 months)
  OS is defined as the time until death due to any cause.
Objective Response Rate (ORR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  ORR is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1.prior to progression or any further therapy.
Disease Control Rate (DCR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD) based on RECIST 1.1.
Quality of Life score (QoL) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  use EORTC QLQ-C30(version 3) questionnaire to evaluate the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong cancer hospital, Jinan, Shandong, China

REFERENCES:
- [Background] Han B, Li K, Zhao Y, Li B, Cheng Y, Zhou J, Lu Y, Shi Y, Wang Z, Jiang L, Luo Y, Zhang Y, Huang C, Li Q, Wu G. Anlotinib as a third-line therapy in patients with refractory advanced non-small-cell lung cancer: a multicentre, randomised phase II trial (ALTER0302). Br J Cancer. 2018 Mar 6;118(5):654-661. doi: 10.1038/bjc.2017.478. Epub 2018 Feb 13. PMID 29438373
- [Result] Syed YY. Anlotinib: First Global Approval. Drugs. 2018 Jul;78(10):1057-1062. doi: 10.1007/s40265-018-0939-x. PMID 29943374
- [Result] Lv Y, Zhang J, Liu F, Song M, Hou Y, Liang N. Targeted therapy with anlotinib for patient with recurrent glioblastoma: A case report and literature review. Medicine (Baltimore). 2019 May;98(22):e15749. doi: 10.1097/MD.0000000000015749. PMID 31145289
- [Result] Shen G, Zheng F, Ren D, Du F, Dong Q, Wang Z, Zhao F, Ahmad R, Zhao J. Anlotinib: a novel multi-targeting tyrosine kinase inhibitor in clinical development. J Hematol Oncol. 2018 Sep 19;11(1):120. doi: 10.1186/s13045-018-0664-7. PMID 30231931